CLINICAL TRIAL: NCT04755868
Title: A Randomized Phase II Clinical Trial of Talazoparib Maintenance Therapy in Triple-negative Breast Cancer Patients Who Showed Platinum-sensitivity on First- or Second-line Platinum-based Chemotherapy
Brief Title: Talazoparib Maintenance Therapy in Triple-negative Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4-2020-1131
Record Dates: First submitted 2021-02-09; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: TNBC - Triple-Negative Breast Cancer
Keywords: BRCA +, Breast cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — talazoparib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maintenance therapy with talazoparib (Experimental): Maintenance therapy with talazoparib (1mg once daily) (once daily 1.0 mg oral administration), 103patients
  Interventions: Drug: Talazoparib
- Maintenance therapy with placebo (Active Comparator): Maintenance therapy with placebo (once daily 1.0 mg oral administration), 103patients
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Talazoparib — The Arm A (Experimental arm) Maintenance therapy with talazoparib (1mg once daily) (once daily 1.0 mg oral administration), 103patients
  Arms: Maintenance therapy with talazoparib
Drug: Placebo — The Arm B (Control arm) Maintenance therapy with placebo (once daily 1.0 mg oral administration), 103patients
  Arms: Maintenance therapy with placebo

SUMMARY:
The investigators propose a randomized phase II clinical trial of talazoparib maintenance therapy in TNBC patients whose tumor showed clinical benefit (platinum-sensitivity) to first- or second-line platinum-based chemotherapy (monotherapy or combination with other agents).

Patients are eligible when they meet at least one of two following platinum-sensitivity criteria:

1. They should have received 6 tri-weekly doses or 18 weekly doses of platinum-based therapy in non-progression status (at least stable disease) at the time of enrollment;
2. They should remain in complete or partial response status after 4-6 tri-weekly doses or 12-18 weekly doses of platinum-based chemotherapy. Eligible patients are enrolled to the trial within 4 to 8 weeks after last chemotherapy and 1:1 randomized to receive talazoparib versus placebo maintenance therapy.

The primary endpoint is PFS by RECIST 1.1 after randomization. The secondary endpoints include OS, time from randomization to second progression or death (PFS2), and objective response rate (ORR) by RECIST 1.1, adverse events by CTCAE 5.0 criteria, quality of life evaluated by EORTC-QLQ-C30, and EuroQoL EQ-5D.

DETAILED DESCRIPTION:
Randomized double-blind placebo controlled phase II trial

This is a double-blind, placebo-controlled randomized phase II study, and the TNBC patients showing platinum-sensitivity after first- or second-line platinum-based chemotherapy will be screened. The total doses of platinum-based chemotherapy will be 4 or 6 doses for tri-weekly regimens and 12 or 18 doses for weekly regimen before randomization

. The platinum sensitivity is determined as follows,

1. Remaining stable disease after 6 tri-weekly doses or 18 weekly doses of platinum-based therapy (stable disease after 6 cycles)
2. Remaining complete or partial response status after 4-6 tri-weekly doses or 12-18 weekly doses of platinum-based chemotherapy (partial or complete response after 4-6 cycles)

The platinum sensitivity of the patients will be determined before enrollment to the clinical trial by review of central investigation institution (Yonsei Cancer Center) based on the the image reading results and, if necessary, the raw imaging data to determine that there is no tumor progression, tumor size increase, or new lesions.

The platinum-based chemotherapy can be either monotherapy or combination doublet chemotherapy of carboplatin or cisplatin with following combination partners: Paclitaxel, Docetaxel, Gemcitabine, Eribulin, Vinorelbine, Capecitabine, and Nab-paclitaxel. The combined targeted therapy agents including bevacizumab will be allowed but should be discontinued before randomization.

The patient with any BRCA1/2 mutation status is eligible. Germline BRCA1/2 test will be performed with reimbursement from South Korean health insurance in the study subject, if the subjects are under the age of 60 or have family history of BRCA-related cancers before enrollment. The testing results will be verified by the investigator. If the germline BRCA1/2 test is not covered by national health insurance (patients over 60 years of age and no family history), the BRCA1/2 germline testing will be performed with study support.

The germline BRCA mutation status will be determined before randomization if the patient do not have BRCA mutation results before. The eligible patients will be assigned to each treatment arm after 1:1 randomization. The patients will be stratified on randomization with following factors.

1. 1st line platinum-based chemotherapy versus 2nd line platinum-based chemotherapy*
2. Response (CR/PR vs. stable disease) to the prior platinum-based chemotherapy
3. BRCA status: wild-type (including benign variants and variants of unknown significance) versus BRCA1/2-mutated (pathogenic mutation)

   * For the patient who recurred within 12 months after the last dose of (neo)adjuvant chemotherapy for operable stage breast cancer, the (neo)adjuvant chemotherapy will be considered as one line of chemotherapy.

The Arm A (Experimental arm) Maintenance therapy with talazoparib (1mg once daily) (once daily 1.0 mg oral administration), 103patients The Arm B (Control arm) Maintenance therapy with placebo (once daily 1.0 mg oral administration), 103patients

The maintenance talazoparib will be initiated 4 to 8 weeks after the last dose of platinum-based chemotherapy. The talazoparib treatment will continue until disease progression by RECIST 1.1, unacceptable toxicity, or death.

Computed tomography or magnetic resonance imaging of the chest, abdomen, and pelvis will be performed at baseline, and every 8 weeks until disease progression after then.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed TNBC patients receiving first- or second-line chemotherapy for recurrent, metastatic, or unresectable disease. The triple-negative breast cancer is defined as ER negative, PR negative, and HER2 negative receptor status

   * ER and PR negative defined as IHC nuclear staining < 1% AND
   * HER2 negative defined as:

     1. IHC 0, 1+ without ISH OR
     2. IHC 2+ and ISH non-amplified (average HER2 gene copy number < 4 signals/cell using single-probe ISH or HER2/CEP17 ratio < 2.0 and average HER2 gene copy number < 4 signals/cell in dual-probe ISH) OR
     3. ISH non-amplified without IHC
2. Female patients with ≥19 years of age
3. Patients on first- or second-line platinum-based (cisplatin or carboplatin) chemotherapy regimen for recurrent, metastatic, or unresectable TNBC showing platinum-sensitivity during chemotherapy

   * The platinum-based chemotherapy can be either monotherapy or combination doublet chemotherapy of carboplatin or cisplatin with following combination partners: Paclitaxel, Docetaxel, Gemcitabine, Eribulin, Vinorelbine, Capecitabine, and Nab-paclitaxel.
   * For the patient who recurred within 12 months after the last dose of (neo)adjuvant chemotherapy for operable stage breast cancer, the (neo)adjuvant chemotherapy will be considered as one line of chemotherapy.
   * The combined targeted therapy agents including bevacizumab will be allowed but should be discontinued before randomization.

   The platinum sensitivity is determined as follows,
   * Remaining stable disease after 6 tri-weekly doses or 18 weekly doses of platinum-based therapy (stable disease after 6 cycles)
   * Remaining complete or partial response status after 4-6 tri-weekly doses or 12-18 weekly doses of platinum-based chemotherapy (partial or complete response after 4-6 cycles)
4. Patients who can receive germline BRCA1/2 mutation test or patients with previously known germline BRCA1/2 mutation status.
5. Provision of informed consent prior to any study specific procedures
6. Measurable disease and/or non-measurable or no evidence of disease assessed at baseline by CT as defined by RECIST 1.1
7. Patients who have received platinum as potentially curative treatment for a prior cancer (eg ovarian cancer) or as adjuvant/neoadjuvant treatment for breast cancer are eligible with at least 12 months elapsed between the last dose of curative platinum-based treatment and initiation of the platinum-based chemotherapy for recurrent, metastatic, or unresectable breast cancer.
8. ECOG performance status 0 or 1
9. Adequate organ function within 14 days before enrollment for treatment A. Absolute neutrophil count (ANC) ≥ 1500 cells/mm3 B. Platelets ≥ 100,000 cells/mm3 C. Hemoglobin ≥ 9.0g/dL with no blood transfusions (packed red blood cells) in the past 7 days D. Bilirubin ≤ 2.0 x ULN E. AST (SGOT) ≤ 3 x ULN (5.0 x ULN if hepatic metastases) F. ALT (SGPT) ≤ 3 x ULN (5.0 x ULN if hepatic metastases) G. Creatinine clearance ≥ 30mL/min as calculated using the Cockcroft-Gault equation or serum creatinine ≤ 1.5 ULN
10. 12-Lead electrocardiogram (ECG) with normal tracing or non-clinically significant changes that do not require medical intervention
11. QTc interval ≤470 msec and without history of Torsades de pointes
12. Not pregnant or nursing, fertile patients must use effective contraception 2 weeks before, during, and for 7 months after completion of study treatment

    * A fertile female patient whose result of the urine test or serum pregnancy test was negative within 72 hours of the first dose. If the test results are positive or not-confirmatory negative, a serum pregnancy test should be performed.
    * The fertile women are required to use proper contraception (inscribed in 11.13 section) during clinical trials and up to seven months after final administration, or agree to be surgically infertile or to stop having heterosexual sex.

    The definition of infertile women is as follows, and the woman who do not fall under this category are judged to be fertile women.
    * Women who have undergone infertility surgery (bilateral tubal resection, bilateral oophorectomy, or uterine resection)
    * Women aged 55 or older who have no natural menstruation for more than 12 months before random assignment
    * Women under the age of 55 with no natural menstruation and a menopause follicle hormone (FSH) concentration of 30 IU/L (or meet the standards of post-menopausal in the local lab) for a period of more than 12 months before randomization
13. No other concurrent severe and/or uncontrolled medical disease which could compromise study participation
14. Adequate treatment washout period before enrollment are below Treatment Washout Period Major surgery ≥ 4 weeks Radiation therapy ≥ 4 weeks (if palliative stereotactic radiation therapy ≥ 2 weeks)
15. For patients with Germline BRCA1/2 mutations, the patients whose use of PARP inhibitors outside this clinical trial after the treatment of the platinum chemotherapy is inappropriate, impossible, or difficult to implement due to the patient's rejection, judged by the investigator or the patient for various reasons (including economic reasons)

Exclusion Criteria:

1. Progression of tumor between start of platinum-based chemotherapy for recurrent, metastatic, or unresectable TNBC and randomization.
2. Severe Cardiac disease (e.g., uncontrolled hypertension, congestive cardiac failure, ventricular arrhythmias, active ischemic heart disease, myocardial infarction within the past year)
3. Current active hepatic or biliary disease (except for Gilbert syndrome, asymptomatic gallstones, liver metastasis or stable chronic liver disease per investigator assessment).
4. Any previous treatment with a PARP inhibitor, including talazoparib
5. Clinically significant uncontrolled medical conditions are not permitted that would limit ability to comply with study procedures, and any other medical condition that places the patient at unacceptable risk of toxicity.
6. Presence of symptomatic CNS metastases or CNS metastases that require local CNS-directed therapy (such as radiotherapy or surgery). Patients with treated brain metastases should be neurologically stable (for 4 weeks post treatment and prior to study enrollment) and without steroid therapy over physiologic dose (> 10mg prednisolone/day) for at least 2 weeks before administration of study drug.
7. Concomitant use of known potent CYP3A4/5 inhibitors such as ketoconazole, itraconazole, ritonavir, indinavir, saquinavir, telithromycin, clarithromycin and nelfinavir.
8. Known active hepatitis B or C infection
9. Significantly altered mental status prohibiting the understanding of the study, or with psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
10. Multiple primary malignancies within 5 years, except adequately resected non-melanoma skin cancer, curatively treated in-situ disease, other solid tumors curatively treated, or contralateral breast cancer.
11. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
12. Patients who are pregnant or nursing, or plan to be pregnant during the scheduled clinical trial period from the screening visit to 7 months after the last administration of the medication.
13. Previous allogeneic bone marrow transplant.
14. Patients with a known hypersensitivity to talazoparib or any of the excipients of the product.
15. Patients who received live-attenuated vaccination with 30 days before the first administration of study drug
16. Unresolved systemic active infection
17. Patients with history of HIV infection

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients with ≥19 years of age
Enrollment: 206 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 months
  Progression-free survival (PFS) after randomization by RECIST 1.1 PFS is defined as time interval from cycle 1 day 1 to tumor progression/death/last follow-up.

SECONDARY OUTCOMES:
Overall survival (OS) | 2 months
  OS is defined as time interval from cycle 1 day 1 to tumor death/last follow-up.
progression-free survival 2 | 2 months
  PFS2 is defined as time interval from cycle 1 day 1 to second tumor progression or death.
Objective response rate | 2 months
  ORR is defined as rate of patients with complete remission (CR) or partial remission (PR) based on RESIST1.1.
Adverse events by CTCAE 5.0 criteria | 2 months
  Safety is based on CTCAE 5.0.
Quality of life (QoL) | 2 months
  Quality of life (QoL) measured by EORTC-QLQ-C30
Progression-free survival(PFS) analysis | 2 months
  Progression-free survival(PFS) analysis using visceral metastasis status as covariate
Quality of life (QoL) | 2 months
  Quality of life (QoL) measured by EuroQoL EQ-5D

CONTACTS AND LOCATIONS:
Overall Officials: Joohyuk sohn, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No